CLINICAL TRIAL: NCT03058042
Title: Outpatient Pelvic Floor Muscle Training Versus Home Pelvic Floor Muscle Training for Stress Urinary Incontinence: Randomized Controlled Trial
Brief Title: Outpatient and Home Pelvic Floor Training for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Fatima Fitz, Physiotherapist, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Urinary Incontinence, Stress
Keywords: Urinary Incontinence, Stress; Pelvic Floor; Exercise; Physical Therapy Modalities
MeSH Terms: conditions — Urinary Incontinence, Stress; Motor Activity

STUDY DESIGN:
Intervention Model Description: Protocol of group I (Outpatient training): Patients will perform 24 outpatient sessions of pelvic floor muscle (PFM) strength training and home training. At the end of one month, the patients will perform PFM evaluation and training progression
  Group II protocol (home training): Patients will perform strength training of the pelvic floor muscles daily at home. At the end of one month, the patients will return for consultation, in which the PFM evaluation and training progression will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home pelvic floor muscle training (Experimental): Patients will perform strength training of the pelvic floor muscles daily at home. The training protocol consists of three sets of 30 slow contractions (type I muscle fibers), with maintenance contraction according to the initial evaluation, followed by three rapid contractions (type II muscle fibers) after each slow contraction. The protocol will account for 90 contractions of the pelvic floor muscles per day. At the end of one month, the patients will return for consultation, in which the MAP evaluation and training progression will be performed.
  Interventions: Other: Exercises of the pelvic floor muscle at home
- Outpatient pelvic floor muscle training (Sham Comparator): The patients will perform 24 outpatient sessions of pelvic floor muscle strength training and home training. The training protocol consists of three sets of 30 slow contractions (type I muscle fibers), with maintenance contraction according to the initial evaluation, followed by three rapid contractions (type II muscle fibers) after each slow contraction. The protocol will account for 90 contractions of the pelvic floor muscles per day. At the end of one month, the patients will perform the evaluation of the MAP and progression of the training.
  Interventions: Other: Exercises of the pelvic floor muscle in the outpatient

INTERVENTIONS:
Other: Exercises of the pelvic floor muscle at home — Patients will perform pelvic floor exercises at home.
  Arms: Home pelvic floor muscle training
Other: Exercises of the pelvic floor muscle in the outpatient — Patients will perform pelvic floor exercises in the outpatient.
  Arms: Outpatient pelvic floor muscle training

SUMMARY:
The objective of this study is to compare the effect of outpatient pelvic floor muscle training versus home pelvic floor muscle training in the treatment of stress urinary incontinence. The hypothesis of this study is that home pelvic floor muscle training is as effective as outpatient pelvic floor muscle training for the treatment of stress urinary incontinence.

DETAILED DESCRIPTION:
Success with the pelvic floor muscle training (PFMT) is hampered by non-adherence, which is related to factors such as inability to contract the pelvic floor muscles and lack of motivation. Thus under supervision by a physiotherapist (outpatient training), PFMT has the potential of improving adherence to training and has been demonstrated to be more effective when compared to unsupervised PFMT (home training). The objective of this study is to compare the effect of outpatient pelvic floor muscle training versus home pelvic floor muscle training in the treatment of stress urinary incontinence. This is a randomized controlled trial and which will be conducted at the Division of Urogynecology and Reconstructive Pelvic Surgery at the Federal University of Sao Paulo, Brazil. As a primary endpoint, the standardized volume test pad (250 mL) will be used. To assert that one of the groups (home PFMT or outpatient PFMT) is superior to the other, it will be necessary to find 38.5% more patients cured when the groups are compared. Secondary outcome measures will be used, assessment of the pelvic floor muscles function, urinary symptoms, quality of life and subjective cure.

ELIGIBILITY:
Inclusion Criteria:

SUI and mixed urinary incontinence with predominant symptoms of SUI with ≥ 2 g of leakage measured by pad test

Exclusion Criteria:

younger than 18 years old chronic degenerative diseases pelvic organ prolapse greater than stage I by POP-Q neurologic or psychiatric diseases inability to contract PFMs previously undergone pelvic floor re-education programs and/or previous pelvic floor surgeries

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Change in pad test | Baseline, after 3 months of treatment
  To quantify the severity of SUI and as the tool to estimate objective cure rate

SECONDARY OUTCOMES:
Change in 7-Day Voiding Diary | Baseline and after 3 months of treatment
  To assess the loss efforts
Change in pelvic floor muscle function (Oxford Grading Scale) | Baseline and after 3 months of treatment
  To assess the function of the pelvic floor muscle
Change in Incontinence Quality-of-Life Questionnaire (I-QoL) | Baseline and after 3 months of treatment
  To quantify the impact of SUI on quality of life
Subjective cure of SUI ("satisfied" or "dissatisfied") | Baseline and after 3 months of treatment
  To evaluate the patient satisfaction with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Castro, Study Director — Universidade Federal de São Paulo
Locations (1):
- Fátima Faní Fitz, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322